CLINICAL TRIAL: NCT00400114
Title: Adjuvant Sutent Following Chemotherapy, Radiation and Surgery For Esophageal Cancer, A Phase II Trial (ASSET)
Brief Title: Sutent Following Chemotherapy, Radiation and Surgery For Resectable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0407-C
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Cancer
Keywords: esophageal; esophagus; cancer; sutent; sunitinib
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Irinotecan; Cisplatin; Radiation; Surgical Procedures, Operative; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sunitinib (Experimental)
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Procedure: Radiation; Procedure: Surgery; Drug: sunitinib (Sutent)

INTERVENTIONS:
Drug: Irinotecan — Irinotecan (50mg/m2)once weekly in weeks 1, 2, 4, 5, 7, and 8
Drug: Cisplatin — Cisplatin (65mg/m2)once weekly in weeks 1, 2, 4, 5, 7, and 8
Procedure: Radiation — Radiation 50 Gy (weeks 4-9)
Procedure: Surgery — Esophagectomy
Drug: sunitinib (Sutent) — sunitinib (Sutent), dose range of 12.5mg - 50mg OD x 1 year post op.

SUMMARY:
The purpose of this study is to see whether or not the combination of cisplatin, irinotecan and radiation, followed by surgery, followed by oral Sutent, is effective and safe for patients with resectable esophageal cancer.

DETAILED DESCRIPTION:
Survival outcomes for resectable esophageal cancer remain poor. Current data strongly support an adjuvant systemic strategy to improve time to progression and survival in this patient population. Adding a well-tolerated oral targeted therapy such as Sutent, after a combined chemo/radiation/surgery approach in this patient population has the potential to impact on the minimal residual disease left behind by relatively effective pre-operative chemoradiation and surgery. This has the potential to improve survival. The primary endpoint is to determine the feasibility and efficacy of adjuvant Sutent therapy (SU11248) after concurrent neoadjuvant therapy with irinotecan, cisplatin, external beam conformal radiotherapy plus surgery for potential resectable esophageal cancer. Preclinical and clinical data suggest that Sutent will have activity in esophageal cancer, as the results of Sutent activity in solid tumors appear to be superior to the results of other antiangiogenic compounds in development for esophageal cancer. Therefore, by extrapolation from promising phase I, II and III Sutent trials we propose to translate the target effects achieved with Sutent to reduce local and systemic therapy failure, and thus metastasis in esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous or adenocarcinoma or the esophagus >20 cm from the incisors, including GE junction tumors (unless of gastric origin).
* Tumors must be technically resectable.
* Clinical T1N1M0, T2-3 N0-1 M0
* Performance status ECOG 0-1
* Medically fit for chemotherapy, radiation and esophagectomy

Exclusion Criteria:

* In situ or clinical T1N0M0, and stage IV (M1a orM1b)
* Cervical esophageal tumors (within 20 cm of the incisors)
* Age <18 or >70
* Participation in another concurrent clinical study involving study drug(s) or treatment with study drug within thirty days prior to the treatment on this study. Concurrent treatment with other experimental drugs or anticancer therapy
* known or suspected drug or alcohol abuse
* Prior treatment for this malignancy except esophageal stenting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09-25 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2016-09-19 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and efficacy of adjuvant Sutent therapy after concurrent neoadjuvant therapy with Irinotecan, Cisplatin, external beam conformal radiotherapy plus surgery for potentially resectable esophageal cancer. | 5 yrs

SECONDARY OUTCOMES:
To assess the impact of adjuvant targeted therapy with Sutent after multimodality therapy for resected esophageal cancer stage II to III, and to compare these data to our current completed trial in the same patient population | 5 yrs
To characterize toxicity of targeted adjuvant therapy with Sutent after multimodality therapy for resected esophageal cancer stage II to III | 2 yrs
To measure time-to-event efficacy variables including: Time to treatment failure and Time to progressive disease | 5 yrs
Survival of patients with esophageal cancer stage II to III with adjuvant targeted therapy added to multimodality treatment protocol | 5 yrs
To determine the pattern of relapse (local versus distant) with the addition of adjuvant targeted therapy to esophageal cancer multimodality therapy | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Knox, MD M.Sc. FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - University Health Network (Princess Margaret & Toronto General Hospitals), Toronto, Ontario

REFERENCES:
- [Background] Horgan AM, Darling G, Wong R, Guindi M, Liu G, Jonker DJ, Lister J, Xu W, MacKay HM, Dinniwell R, Kim J, Pierre A, Shargall Y, Asmis TR, Agboola O, Seely AJ, Ringash J, Wells J, Marginean EC, Haider M, Knox JJ. Adjuvant sunitinib following chemoradiotherapy and surgery for locally advanced esophageal cancer: a phase II trial. Dis Esophagus. 2016 Nov;29(8):1152-1158. doi: 10.1111/dote.12444. Epub 2015 Dec 10. PMID 26663741